CLINICAL TRIAL: NCT06751706
Title: Detection of Mycobacterium Tuberculosis in Blood of TB Patients and Their Contacts in Uganda
Acronym: MICRO-LTBI_UG
Status: Enrolling by invitation | Type: Observational
Sponsor: Queen Mary University of London (Other)
Collaborators: Makerere University (Other)
Responsible Party: Sponsor
Other Study IDs: IDI-REC-2023-80
Record Dates: First submitted 2024-12-20; First posted 2024-12-30 (Actual); Last update posted 2025-06-08 (Actual); Status verified 2025-06

CONDITIONS: Tuberculosis; Latent Tuberculosis
Keywords: Tuberculosis; Latent tuberculosis; TB; TB Infection; TB Biomarker; Blood test for TB
MeSH Terms: conditions — Tuberculosis; Latent Tuberculosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Peripheral blood mononuclear cells
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- Group A: TB patients: New diagnosis of smear-positive or Xpert-confirmed pulmonary TB
- Group B: Recent TB contacts: Household contact with an index case of smear-positive pulmonary TB recruited to Group A.
- Group C: Historical TB contacts: Participant in previous TB household contact study

SUMMARY:
Mycobacterium tuberculosis (Mtb) is a major human pathogen, responsible for an estimated 10.6 million cases of active tuberculosis (TB) and 1.6 million deaths in 2021. Most adult cases of active TB arise from progression of latent tuberculosis infection (LTBI), whose global prevalence is estimated at 23%. Preventive therapy (e.g. a 6-month course of the anti-TB drug isoniazid) is effective in reducing risk of progression from LTBI to active TB. Global roll-out of preventive therapy will be required to achieve the World Health Organization target of TB elimination by 2050, but this will only be cost-effective and implementable if targeted at the 10-20% of latently infected individuals who are at highest risk of disease progression.

There is currently no gold standard test for LTBI. Existing diagnostic - the tuberculin skin test (TST) and Interferon-γ Release Assays (IGRA) - diagnose Mtb infection by detecting memory T cell responses to Mtb antigens. Their value is limited by very low positive predictive value (PPV) for progression to active TB (1.5% for TST, 2.7% for IGRA), inability to detect antimicrobial resistance in latently infected individuals and lack of response to administration of preventive therapy. Development of a nucleic acid amplification test (NAAT) for LTBI could overcome these limitations by allowing targeting of preventive therapy at latently infected individuals with the highest risk of progression to active TB, with antimicrobial selection guided by genetic antimicrobial resistance profiling and capacity for test of cure on treatment completion.

DETAILED DESCRIPTION:
For many years, development of such a test was not considered realistic due to the paucibacillary nature of LTBI and uncertainty regarding the cellular location of Mtb bacilli in LTBI. However, the investigators and others have recently reported that Mtb DNA can be detected in the peripheral blood of latently infected TB contacts in both high- and low-burden settings. In our studies, which utilized digital polymerase chain reaction (dPCR) to detect Mtb DNA in peripheral blood mononuclear cell (PBMC) subsets of TB contacts in Ethiopia, signal was detected more frequently in extracts of CD34+ PBMC (hematopoietic stem cells [HSC] and their progenitors) vs. CD34- PBMC, but it was not restricted to them. Administration of isoniazid preventive therapy (IPT) reduced the proportion of participants in whom Mtb DNA could be detected in PBMC, showing that this signal is dynamic and suggesting that presence of Mtb DNA may reflect presence of viable bacilli. The investigatorsalso sequenced Mtb DNA in PBMC extracts using targeted next-generation sequencing (tNGS) to reveal mutations that confer antimicrobial drug resistance.

These exciting results demonstrate the potential for development of a NAAT for detection and genomic drug-resistance testing of LTBI in peripheral blood. However, questions remain regarding whether detection of Mtb DNA in the blood of symptomatic individuals associates with the ability to visualize or culture bacilli in blood, which has been done in patients with active TB. Moreover, our existing method for detection of Mtb DNA in CD34+ PBMC using dPCR is not currently suitable for field use, as samples require lengthy laboratory processing. The GeneXpert platform, which can give results in less than 2 hours, has previously been used to detect Mtb DNA in whole blood of HIV-infected patients with active TB. Sensitivity of the Xpert® MTB/RIF Ultra assay (Xpert Ultra, which has a limit of detection [LOD] of 15.6 colony-forming units [CFU]/ml versus 112.6 CFU/ml for the original Xpert® MTB/RIF [assay) is sufficient to detect Mtb DNA in the range demonstrated in blood of latently infected TB contacts in Ethiopia and Uganda (20 to 1000 copies of rpoB in the majority of Mtb DNA-positive individuals). However, detection of Mtb in blood of latently infected individuals has not previously been attempted using this platform. Finally, the investigators wish to expand knowledge by comparing detection of Mtb DNA in recent vs. historical TB contacts, and by including patients with active TB as a positive control group.

The investigators therefore propose to conduct a study to compare the sensitivity of different methodologies for detection of Mtb and genomic drug resistance in peripheral blood of TB patients and recently vs. remotely exposed asymptomatic TB contacts in Kampala, Uganda.

Study objectives Primary objective

The primary objective of this study is to determine whether Mycobacterium tuberculosis (Mtb) can be detected in the blood of recent TB contacts, recruited in Kampala, Uganda, using any of the following methods:

* Digital PCR
* GeneXpert® MTB/RIF Ultra (Cepheid)
* Fluorescence microscopy
* Blood culture
* Targeted Next-Generation Sequencing

Secondary objectives

Secondary objectives of this study are:

1. To determine whether Mtb persists in the blood of remotely exposed (historical) TB contacts, recruited in the same setting, and using the same methods.
2. To determine whether Mtb can be detected in the blood of patients with newly-diagnosed active TB, recruited in the same setting, and using the same methods.
3. To establish whether detection of Mtb in blood using the methods above associates with any of the following biomarkers of host immune response:

   * QFT-Plus
   * Blood RNA signatures for incipient tuberculosis
   * Antibody profiles
4. To determine whether Mtb strains isolated from the sputum/blood of index cases with pulmonary TB are genetically identical to those detected in the blood of their recent contacts.

Primary endpoint Proportion of TB patients and their contacts in whom Mtb DNA can be detected in peripheral blood using digital PCR.

Secondary endpoints

1. Proportion of TB patients and their contacts in whom Mtb DNA can be detected in peripheral blood using the following methods:

   * GeneXpert® MTB/RIF Ultra (Cepheid)
   * Fluorescence microscopy
   * Blood culture
   * Targeted Next-Generation Sequencing
2. Proportion of TB patients and their contacts with positive results for either of the following assays:

   * QFT-Plus
   * Blood RNA signatures for incipient tuberculosis
   * Antibody profiles
3. Genetic sequences of Mtb strains isolated from the sputum/blood of index cases with pulmonary TB and blood of these participants and their asymptomatic household contacts.

ELIGIBILITY:
TB patients (Group A):

Inclusion Criteria:

* Able and willing to give written informed consent to participate
* Age ≥18 years
* New diagnosis of smear-positive or Xpert-confirmed pulmonary TB
* At least one asymptomatic adult household contact likely to fulfil TB contact eligibility criteria below

Exclusion criteria:

* More than 7 days of anti-TB treatment taken
* Confirmed or suspected pregnancy (female participants)
* Existing medical condition which in the opinion of the investigator may adversely affect the participant's safety or ability to participate in the study.

Recent TB contacts (Group B):

Inclusion Criteria:

* Able and willing to give written informed consent to participate
* Age ≥18 years
* Household contact with an index case of smear-positive pulmonary TB in Group A above.

Exclusion Criteria:

* Clinical or radiological features of active TB
* Current or previous anti-TB treatment
* Confirmed or suspected pregnancy (female participants)
* Existing medical condition which in the opinion of the investigator may adversely affect the participant's safety or ability to participate in the study.

Historical TB contacts (Group C):

Inclusion Criteria:

* Able and willing to give written informed consent to participate
* Age ≥18 years
* Participant in previous TB household contact study

Exclusion Criteria:

* Clinical or radiological features of active TB
* Current or previous anti-TB treatment
* Confirmed or suspected pregnancy (female participants)
* Existing medical condition which in the opinion of the investigator may adversely affect the participant's safety or ability to participate in the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: * 20 index cases of pulmonary TB (Group A)
  * 20 recent household contacts of Group A index cases
  * 20 historical TB contacts who previously participated in a TB household contact study
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2024-09-30 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-04-30 (Estimated)

PRIMARY OUTCOMES:
Mtb DNA prevalence | 1 year
  Prevalence of detectable Mtb in each group

SECONDARY OUTCOMES:
Mtb detection using alternative methods | 1 year
  Determine if Mtb can be detected in the blood of TB patients and their contacts, recruited in Kampala, Uganda, using any of the following methods:
  * GeneXpert® MTB/RIF Ultra (Cepheid)
  * Fluorescence microscopy
  * Blood culture
  * Targeted Next-Generation Sequencing
Mtb DNA detection association with IGRA and RNA signatures for incipient TB | 1 year
  Mtb DNA detection in blood and association with any of the following biomarkers of host immune response:
  * QFT-Plus
  * Blood RNA signatures for incipient tuberculosis
Strain correlation between index case and contact | 1 year
  To determine if Mtb strains isolated from the sputum of index cases with pulmonary TB are genetically identical to those detected in the blood of their contacts.

CONTACTS AND LOCATIONS:
Overall Officials: Adrian Martineau, PhD, Principal Investigator — Queen Mary University London
Locations (1):
- Infectious diseases institute, Makarere University, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: Undecided